CLINICAL TRIAL: NCT00686998
Title: A Phase IIa, Double-blind, Double-Dummy, Placebo-controlled, Randomized, Parallel-Group Study to Assess the Efficacy, Safety, Tolerability, and Pharmacokinetics of AZD2624 in Adult Schizophrenia Patients
Brief Title: Phase IIA Study in Patients With Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D0970C00004
Record Dates: First submitted 2008-05-28; First posted 2008-05-30 (Estimated); Results first posted 2011-06-23 (Estimated); Last update posted 2013-03-29 (Estimated); Status verified 2013-03

CONDITIONS: Schizophrenia
Keywords: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — 3-((methylsulfonyl)amino)-2-phenyl-N-(1-phenylpropyl)quinolin-4-carboxamide; Olanzapine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- AZD2624 (Experimental): AZD2624 40 mg
  Interventions: Drug: AZD2624
- Olanzapine (Other): Olanzapine 15 mg
  Interventions: Drug: Olanzapine
- Placebo (Placebo Comparator): Matching Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD2624 — Oral Suspension
  Arms: AZD2624
Drug: Olanzapine — PO BID
  Other Names: Zyprexa
  Arms: Olanzapine
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study is designed to assess the effects of AZD 2624 in patients with schizophrenia

ELIGIBILITY:
Inclusion Criteria:

* Females of non-childbearing potential
* Diagnosis of Schizophrenia

Exclusion Criteria:

* Clinically relevant disease and /or abnormalities.
* Alcohol or substance abuse not in remission
* Enrollment in another investigational study within 30 days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2008-05; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dhaval Desai, MD, Study Director — AstraZeneca
Locations (1):
- Research Site, Rockville, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 2 centers in the US were initiated and enrolled patients. 159 patients enrolled, of which 106 randomized
Pre-assignment Details: Patients were screened up to 21 days, and admitted to the Clinical Research Unit (CRU) for a maximum of 2 days until eligibility was determined. Once eligibility was determined, patients currently on medication entered a 7 days washout period, patients not currently on medication had a 3 day washout, prior to randomization to study medication.
Period: Overall Study
Arm/Group | AZD2624 | Placebo | Olanzapine
Started | 43 (Randomized & received study medication) | 41 (Randomized & received study medication) | 22 (Randomized & received study medication)
Randomized | 43 | 41 | 22
Received Treatment | 43 | 41 | 22
Eligible for Efficacy Analysis | 42 | 39 | 21
Completed Scheduled Treatment | 30 | 33 | 18
Completed | 30 | 33 | 18
Not Completed | 13 | 8 | 4
Not completed — Adverse Event | 3 | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1 | 2
Not completed — Lack of Efficacy | 7 | 5 | 0
Not completed — Other | 0 | 0 | 1
Not completed — Safety Reasons | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD2624 | Placebo | Olanzapine | Total
Number analyzed (Participants) | 43 | 41 | 22 | 106
Age Continuous [Mean (Standard Deviation); unit: Year] | 40.1 (12) | 40.2 (11.6) | 35.3 (8.7) | 39.2 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 0 | 5
  Male | 40 | 39 | 22 | 101

OUTCOME MEASURES:

1. Primary Outcome: Positive and Negative Syndrome Scale (PANSS) Total Score Change From Baseline
Description: PANSS total score, sum of 30 item scores (each on a 0 to 7 scale), assesses positive and negative symptoms of psychopathology on a continuous scale from 0 (the best) to 210 (the worst). Day 28 value was calculated using last observation carried forward (LOCF). Change from baseline was calculated as Day 28 value minus baseline value.
Time Frame: Baseline, Day 28
Measure: Mean (Standard Error); unit: Points on a scale
Groups:
- Placebo: Placebo
Arm/Group | AZD2624 | Placebo | Olanzapine
Number analyzed (Participants) | 42 | 39 | 21
Points on a scale | 1.40 (2.27) | 4.51 (2.35) | -8.79 (3.2)

ADVERSE EVENTS:
Arm/Group | AZD2624 | Placebo | Olanzapine
Serious Adverse Events (participants affected / at risk) | 4/43 | 2/41 | 0/22
Other Adverse Events (participants affected / at risk) | 29/43 | 27/41 | 18/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AZD2624 (N=43) | Placebo (N=41) | Olanzapine (N=22)
Psychotic disorder (Psychiatric disorders) | 4 | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AZD2624 (N=43) | Placebo (N=41) | Olanzapine (N=22)
Headache (Nervous system disorders) | 7 | 0 | 3
Weight Increased (Investigations) | 0 | 0 | 9
Sedation (Nervous system disorders) | 4 | 1 | 3
Somnolence (Nervous system disorders) | 3 | 1 | 4
Vomiting (Gastrointestinal disorders) | 6 | 1 | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 5 | 1
Nausea (Gastrointestinal disorders) | 5 | 1 | 1
Psychotic Disorder (Psychiatric disorders) | 4 | 3 | 0
Constipation (Gastrointestinal disorders) | 1 | 4 | 1
Dizziness (Nervous system disorders) | 1 | 4 | 0
Increased Appetite (Metabolism and nutrition disorders) | 0 | 1 | 4
Stomach Discomfort (Gastrointestinal disorders) | 2 | 3 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 3 | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0
Dry Mouth (Gastrointestinal disorders) | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days